CLINICAL TRIAL: NCT02798211
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Safety and Efficacy of Secukinumab 300 mg and 150 mg in Adult Patients With Active Psoriatic Arthritis After 16 Weeks of Treatment Compared to Placebo and to Assess the Safety, Tolerability and Efficacy up to 52 Weeks
Brief Title: Study to Evaluate the Safety and Efficacy of Secukinumab 300 mg and 150 mg in Adult Patients With Active Psoriatic Arthritis (PsA) After 16 Weeks of Treatment Compared to Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457FUS01
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Psoriatic Arthritis
Keywords: PsA; ACR; CASPAR; inflammatory arthritis; spondylitis
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis; Spondylitis | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: Study design displays results combined as two or more Arms/Groups. Patients assigned to Placebo arm in Treatment Period 1 (TP1) may have switched to Secukinumab 300mg in Treatment Period 2 (TP2). Summaries by group were performed cumulatively by actual treatment received (as follows) for every visit until Week 16 groups in Treatment Period 1: · Secukinumab 300mg (Group 1) · Secukinumab 150mg (Group 2) · Placebo (Group 3) For entire treatment period, summaries by treatment group were performed cumulatively by the actual treatment received (as follows) for every visit til Week 52, including patients who switched at Weeks 16, 28, 40. For safety variables · Any Secukinumab 150 mg (Group 2) · Any Secukinumab 300mg (Group 1) · Any Secukinumab (Group 3) Hence, participants who received "Placebo" in TP1 were combined with participants who received "Any Secukinumab" in "Group 3" and "Any Secukinumab 300mg" in "Group 1" in TP2. Safety is presented for the ENTIRE period, including TP1 and TP2
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): secukinumab 300mg s.c. injection
  Interventions: Drug: Secukinumab 300 mg
- Group 2 (Active Comparator): secukinumab 150 mg s.c. injection
  Interventions: Drug: Secukinumab 150 mg
- Group 3 (Placebo Comparator): Placebo s.c. injection
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Secukinumab 300 mg — 150 mg x 2 s.c. injection
  Other Names: AIN457
  Arms: Group 1
Drug: Secukinumab 150 mg — 150 mg s.c. injection
  Other Names: AIN457
  Arms: Group 2
Other: Placebo — Placebo
  Other Names: s.c. injection
  Arms: Group 3

SUMMARY:
To demonstrate that the efficacy of secukinumab 300 mg at Week 16 was superior to placebo in adult patients with active PsA based on the proportion of patients achieving an American College of Rheumatology 20 (ACR20) response.

DETAILED DESCRIPTION:
Treatment Period 1 was defined as the period from Randomization through Week 16 (prior to the Week 16 dose). At the start of placebo-controlled Treatment Period 1, patients were randomized via Interactive Response Technology (IRT) in a 2:2:1 ratio to 1 of 3 treatment groups.

Group 1- Secukinumab 300 mg: secukinumab 300 mg (2 s.c. injections of the 150-mg dose) once weekly for 5 weeks (at Baseline, Weeks 1, 2, 3, and 4), followed by dosing every 4 weeks.

Group 2- Secukinumab 150 mg: secukinumab 150 mg (1 s.c. injection of the 150-mg dose and 1 s.c. injection of placebo) once weekly for 5 weeks (at Baseline, Weeks 1, 2, 3, and 4), followed by dosing every 4 weeks.

Group 3- Placebo: placebo (2 s.c. injections of 150 mg secukinumab placebo per dose) once per week for 5 weeks (at Baseline, Weeks 1, 2, 3, and 4), followed by dosing every 4 weeks.

At each study treatment visit 2 s.c. injections in the form of prefilled syringes (PFS) were administered. This was necessary to maintain the blind, as secukinumab in PFS is available in either 1.0 mL (150 mg) or 2 x 1.0 mL (300 mg). Placebo to secukinumab was also available in 1.0 mL to match the active drug.

Rescue medication was not allowed before completion of Week 16 assessments.

Treatment Period 2 patients receiving secukinumab 300 mg (Group 1) continued to receive the same dose up to Week 48.

At Weeks 16, 28, and 40 patients on secukinumab 150 mg (Group 2) were classified as responders (≥20% improvement from BL in both tender and swollen joint counts) or nonresponders.

* At Weeks 16, 28, and 40 patients on secukinumab 150 mg (Group 2) who were responders continued to receive secukinumab 150 mg (1.0 mL) plus placebo (1.0 mL) every 4 weeks until next evaluation of responder status at Weeks 28 or 40.
* Patients who did not meet the responder criteria at Week 16, 28, or 40 started receiving secukinumab 300 mg s.c. every 4 weeks and continued this dose up to Week 48.
* Patients on placebo (Group 3) regardless of their responder status started receiving secukinumab 300 mg s.c. every 4 weeks from Week 16 up to Week 48.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female patients at least 18 years of age
* Diagnosis of PsA classified by CASPAR criteria and with symptoms for at least 6 months with moderate to severe PsA who must have at Baseline ≥3 tender joints out of 78 and ≥3 swollen out of 76 (dactylitis of a digit counts as one joint each)
* Rheumatoid factor and/or anti-CCP antibodies negative at screening
* A target skin psoriatic lesion and a PASI score of 1 or greater

Exclusion Criteria:

* Chest X-ray with evidence of ongoing infectious or malignant process
* Patients who ever received biologic immunomodulating agents including those targeting TNFα, IL-6 and IL-12/23 investigational or approved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (55):
- United States (54):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, El Cajon, California
  - Novartis Investigative Site, Fountain Valley, California
  - Novartis Investigative Site, La Jolla, California
  - Novartis Investigative Site, La Mesa, California
  - Novartis Investigative Site, Upland, California
  - Novartis Investigative Site, Aventura, Florida
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, DeBary, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, North Naples, Florida
  - Novartis Investigative Site, Palm Harbor, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Plantation, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Duluth, Georgia
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Worcester, Massachusetts
  - Novartis Investigative Site, Battle Creek, Michigan
  - Novartis Investigative Site, Kalamazoo, Michigan
  - Novartis Investigative Site, Eagan, Minnesota
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Ridgewood, New Jersey
  - Novartis Investigative Site, Summit, New Jersey
  - Novartis Investigative Site, Albany, New York
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, Lake Success, New York
  - Novartis Investigative Site, Orchard Park, New York
  - Novartis Investigative Site, Potsdam, New York
  - Novartis Investigative Site, Saranac Lake, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, New Bern, North Carolina
  - Novartis Investigative Site, Marion, Ohio
  - Novartis Investigative Site, Perrysburg, Ohio
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Orangeburg, South Carolina
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Mesquite, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Spokane, Washington
- Novartis Investigative Site, Santurce, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Nguyen T, Churchill M, Levin R, Valenzuela G, Merola JF, Ogdie A, Orbai AM, Scher JU, Kavanaugh A, Kianifard F, Rollins C, Calheiros R, Chambenoit O. Secukinumab in United States Biologic-Naive Patients With Psoriatic Arthritis: Results From the Randomized, Placebo-Controlled CHOICE Study. J Rheumatol. 2022 Aug;49(8):894-902. doi: 10.3899/jrheum.210912. Epub 2022 Apr 15. PMID 35428722
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=340

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 349 patients screened for the study, 271 passed screening and 258 were randomized (103 to secukinumab 300 mg, 103 to secukinumab 150 mg, and 52 to placebo). A higher percentage of patients in the secukinumab 300 mg group completed Period 1 (94.2%) than in the secukinumab 150 mg (90.3%) or placebo (88.5%) groups.
Pre-assignment Details: This was a 2-Period study in which participants were randomized to one of three treatment groups (i.e., "secukinumab 300mg s.c. injection", "secukinumab 1500mg s.c. injection" and "placebo s.c. injection") in Period 1 and then some participants switched to Arms/Groups "Group 4", "Group 5", and "Group 6", in Period 2.
Groups:
- Group 4: Secukinumab 150 mg - 150 mg (R)
- Group 5: Secukinumab 150 mg - 300 mg (NR)
- Group 6: Placebo - Secukinumab 300 mg
Period: Period 1
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Started (Screened patients=349 Screen passed patient=271 Screened failure=78 Randomized=103) | 103 | 103 | 52 | 0 | 0 | 0
Completed | 97 | 93 | 46 | 0 | 0 | 0
Not Completed | 6 | 10 | 6 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal of Informed Consent | 2 | 7 | 3 | 0 | 0 | 0
Period: Period 2
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Started (Completed treatment period 1 and continued to treatment period 2) | 97 | 0 | 0 | 50 | 42 | 46
Completed (Completed treatment period 2) | 83 | 0 | 0 | 43 | 34 | 40
Not Completed | 14 | 0 | 0 | 7 | 8 | 6
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 2 | 2
Not completed — Adverse Event | 5 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Technical problems | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal of Informed Consent | 1 | 0 | 0 | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Randomized Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 103 | 103 | 52 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (12.56) | 51.3 (14.58) | 53.1 (12.67) | 52.2 (80.86)
Age, Customized [Count of Participants; unit: Participants]
  ≥18-<40 | 20 | 20 | 8 | 48
  ≥40-<65 | 65 | 61 | 35 | 161
  ≥65-<75 | 14 | 18 | 9 | 41
  ≥75 | 4 | 4 | 0 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 47 | 29 | 126
  Male | 53 | 56 | 23 | 132
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 9 | 10 | 1 | 20
  Black | 2 | 2 | 3 | 7
  Caucasian | 88 | 88 | 45 | 221
  Native American | 0 | 1 | 1 | 2
  Other | 2 | 0 | 2 | 4
  Pacific Islander | 1 | 1 | 0 | 2
  Unknown | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Achieving American College of Rheumatology Score of at Least 20% (ACR20) Response Criteria on Secukinumab 300 mg and 150 mg vs. Placebo at Week 16
Description: A patient was considered as improved according to the ACR20 criteria if she/he had at least 20% improvement in two of the following measures:Tender joint count, Swollen joint count and at least 3 of the following 5 measures: Patient's assessment of pain, Patient's global assessment disease activity, Physician's global assessment of disease activity, Health Assessment Questionnaire (HAQ©) score,Acute phase reactant (hsCRP or ESR).
  Odds ratio, 95% confidence interval for odds ratio, and p-value are from a logistic regression model with treatment (3 treatment groups), methotrexate usage at baseline (yes, no) and body weight (kg) as explanatory variables.
Time Frame: 16 Weeks
Population: The Full Analysis Set (FAS) includes all patients assigned study medication. Patients inappropriately randomized (e.g., IRT was called in error for randomization of a screen failed patient) were excluded from analysis set. Following the intent-to-treat principle, patients were analyzed according to the treatment they were assigned at randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 103 | 103 | 52
percentage of participants | 51.46 | 36.89 | 23.08
Statistical Analysis 1: Comparison: Group 1 vs Group 2; secukinumab 300mg s.c. injection, 16 weeks; Test type: Superiority; p = 0.0011, Regression, Logistic; Statistical analysis (logistic regression) of ACR20 response in treatment period 1 (non-responder imputation); Odds Ratio (OR) = 3.51, 95% CI 2-sided [1.65 to 7.45]
Statistical Analysis 2: Comparison: Group 2; secukinumab 150 mg s.c. injection, 16 weeks; Test type: Superiority; p = 0.0961, Regression, Logistic; Statistical analysis (logistic regression) of ACR20 response in treatment period 1 (non-responder imputation); Odds Ratio (OR) = 1.92, 95% CI 2-sided [0.89 to 4.15]

2. Secondary Outcome: Percentage of Patients With Dactylitis in the Subset of Subjects Who Have Dactylitis at Week 16
Description: The percent of patients in the Dactylitis Subset with dactylitis in the secukinumab 300 mg group at Week 16. Dactylitis is severe inflammation of the finger and toe joints.
  Odds ratio, 95% confidence interval for odds ratio, and p-value are from a logistic regression model with treatment (3 treatment groups), methotrexate usage at baseline (yes, no) and body weight (kg) as explanatory variables.
Time Frame: Week 16
Population: Dactylitis Subset: The Dactylitis Subset comprises patients who have LDI >= 1 at baseline
Measure: Number; unit: percent of participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 49 | 52 | 23
percent of participants | 53.06 | 44.23 | 65.22
Statistical Analysis 1: Comparison: Group 1; secukinumab 300 mg s.c. injection, 16 weeks; Test type: Superiority; p = 0.3330, Regression, Logistic; Statistical analysis (logistic regression) of presence of dactylitis by visit in treatment period 1 (non-responder imputation); Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.22 to 1.68]
Statistical Analysis 2: Comparison: Group 2; secukinumab 150 mg s.c. injection, 16 weeks; Test type: Superiority; p = 0.0841, Regression, Logistic; Statistical analysis (logistic regression) of presence of dactylitis in treatment period 1 (non-responder imputation); Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.14 to 1.13]

3. Secondary Outcome: Percentage of Patients With Enthesitis in the Subset of Subjects Who Have Enthesitis at Baseline (SPARCC) at Week 16
Description: Enthesitis, also called enthesopathy, is inflammation of the entheses, the sites where tendons or ligaments insert into the bone.
  Odds ratio, 95% confidence interval for odds ratio, and p-value are from a logistic regression model with treatment (3 treatment groups), methotrexate usage at baseline (yes, no) and body weight (kg) as explanatory variables.
Time Frame: 16 Weeks
Population: Spondyloarthritis Research Consortium of Canada Enthesitis Index (SPARCC) subset. The SPARCC Subset is comprised of patients who have SPARCC >= 1 at baseline. Score range is 0-16 sites where a higher indicates more enthesitis.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 72 | 76 | 39
percentage of participants | 63.89 | 57.89 | 76.92
Statistical Analysis 1: Comparison: Group 1; secukinumab 300mg s.c. injection, 16 weeks; Test type: Superiority; p = 0.1618, Regression, Logistic; Statistical analysis (logistic regression) of presence of enthesitis (SPARCC) in treatment period 1 (non-responder imputation); Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.21 to 1.30]
Statistical Analysis 2: Comparison: Group 2; secukinumab 150mg s.c. injection, 16 weeks; Test type: Superiority; p = 0.0898, Regression, Logistic; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.19 to 1.13]

4. Secondary Outcome: Percentage of Patients With Enthesitis in the Subset of Subjects Who Have Enthesitis at Week 16 (LEI)
Description: Enthesitis, also called enthesopathy, is inflammation of the entheses, the sites where tendons or ligaments insert into the bone.
  LEI=Leeds Enthesitis Index
Time Frame: 16 Weeks
Population: LEI subset: The LEI Subset comprises patients who have LEI >= 1 at baseline. LEI uses 6 sites for evaluation of enthesitis, so the range is 0-6 withy a higher number indicating more arthritis.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 66 | 67 | 34
percentage of participants | 56.06 | 52.24 | 82.35
Statistical Analysis 1: Comparison: Group 1; secukinumab 300mg s.c. injection, 16 weeks; Test type: Superiority; p = 0.0125, Regression, Logistic; Statistical analysis (logistic regression) of presence of enthesitis (LEI) in treatment period 1 (non-responder imputation); Odds Ratio (OR) = 0.27, 95% CI 2-sided [0.09 to 0.75]
Statistical Analysis 2: Comparison: Group 2; secukinumab 150mg s.c. injection, 16 weeks; Test type: Superiority; p = 0.0086, Regression, Logistic; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.25, 95% CI 2-sided [0.09 to 0.70]

5. Secondary Outcome: Percentage of Patients With Enthesitis in the Subset of Subjects Who Have Enthesitis at Week 16 (Combined SPARCC and LEI)
Description: Statistical analysis (logistic regression) of presence of enthesitis (Combined SPARCC and LEI) by visit - in treatment period 1 (non-responder imputation) (Combined SPARCC and LEI Subset)
  Enthesitis, also called enthesopathy, is inflammation of the entheses, the sites where tendons or ligaments insert into the bone.
  Odds ratio, 95% confidence interval for odds ratio, and p-value are from a logistic regression model with treatment (3 treatment groups), methotrexate usage at baseline (yes, no) and body weight (kg) as explanatory variables.
Time Frame: 16 Weeks
Population: Combined SPARCC and LEI Subset: The LEI and SPARCC Subset comprises patients who have an enthesitis score >= 1 when sites from LEI and SPARCC are assessed together at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 74 | 76 | 39
percentage of participants | 62.16 | 59.21 | 82.05
Statistical Analysis 1: Comparison: Group 1; secukinumab 300mg s.c. injection, 16 weeks; Test type: Superiority; p = 0.0338, Regression, Logistic; Statistical analysis (logistic regression) of presence of enthesitis (SPARCC and LEI) in treatment period 1 (non-responder imputation); Odds Ratio (OR) = 0.35, 95% CI 2-sided [0.13 to 0.92]
Statistical Analysis 2: Comparison: Group 2; secukinumab 150mg s.c. injection, 16 weeks; Test type: Superiority; p = 0.0359, Regression, Logistic; [statistical method as in outcome 5, analysis 1]; Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.14 to 0.93]

6. Secondary Outcome: Percentage of Patients Achieving ACR50 Response Criteria on Secukinumab 300 or 150 mg vs. Placebo at Week 16
Description: A patient was considered as improved according the ACR50 criteria if she/he had at least 50% improvement in the two of the following measures: Tender joint count, Swollen joint count and at least 3 of the following 5 measures: Patient's assessment of pain, Patient's global assessment disease activity,Physician's global assessment of disease activity, Health Assessment Questionnaire (HAQ©) score,Acute phase reactant (hsCRP or ESR)
  Statistical analysis (logistic regression) of ACR50 response by visit - in treatment period 1 (non-responder imputation) (Full Analysis Set)
  Odds ratio, 95% confidence interval for odds ratio, and p-value are from a logistic regression model with treatment (3 treatment groups), methotrexate usage at baseline (yes, no) and body weight (kg) as explanatory variables.
Time Frame: 16 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 103 | 103 | 3
percentage of participants | 28.16 | 24.27 | 5.77
Statistical Analysis 1: Comparison: Group 1; secukinumab 300mg s.c. injection, week 16; Test type: Superiority; p = 0.0038, Regression, Logistic; Statistical analysis (logistic regression) of ACR50 response in treatment period 1 (non-responder imputation); Odds Ratio, log = 6.30, 95% CI 2-sided [1.81 to 21.88]
Statistical Analysis 2: Comparison: Group 2; secukinumab 150 mg s.c. injection, week 16; Test type: Superiority; p = 0.0149, Regression, Logistic; Statistical analysis (logistic regression) of ACR50 response by visit in treatment period 1 (non-responder imputation); Odds Ratio (OR) = 4.77, 95% CI 2-sided [1.36 to 16.77]

7. Secondary Outcome: Percentage of Patients Achieving ACR70 Response Criteria on Secukinumab 300 or 150 mg vs. Placebo at Week 16
Description: A patient was considered as improved according the ACR70 criteria if she/he had at least 70% improvement in the two of the following measures: Tender joint count, Swollen joint count and at least 3 of the following 5 measures: Patient's assessment of pain, Patient's global assessment disease activity,Physician's global assessment of disease activity, Health Assessment Questionnaire (HAQ©) score,Acute phase reactant (hsCRP or ESR)
  Statistical analysis (logistic regression) of ACR70 response by visit - in treatment period 1 (non-responder imputation)
  Odds ratio, 95% confidence interval for odds ratio, and p-value are from a logistic regression model with treatment (3 treatment groups), methotrexate usage at baseline (yes, no) and body weight (kg) as explanatory variables.
Time Frame: 16 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 103 | 103 | 52
percentage of participants | 17.48 | 10.68 | 1.92
Statistical Analysis 1: Comparison: Group 1; secukinumab 300mg s.c. injection, week 16; Test type: Superiority; p = 0.0243, Regression, Logistic; Statistical analysis (logistic regression) of ACR70 response in treatment period 1 (non-responder imputation); Odds Ratio, log = 10.50, 95% CI 2-sided [1.36 to 81.30]
Statistical Analysis 2: Comparison: Group 2; secukinumab 150 mg s.c. injection, week 16; Test type: Superiority; p = 0.1120, Regression, Logistic; Statistical analysis (logistic regression) of ACR70 response by visit in treatment period 1 (non-responder imputation); Odds Ratio (OR) = 5.42, 95% CI 2-sided [0.67 to 43.64]

8. Secondary Outcome: Percentage of Patients Achieving a PASI75 Response in the Subgroup of Subjects Who Have ≥3% Skin Involvement With Psoriasis at Week 16
Description: A 75% reduction in the Psoriasis Area and Severity Index (PASI) score (PASI 75) is above the current benchmark of primary endpoints for most clinical trials with endpoints of psoriasis.
Time Frame: 16 Weeks
Population: Psoriasis Subset: The psoriasis subset comprises patients having Body Surface Area (BSA) >= 3% at baseline
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 79 | 83 | 43
percentage of participants | 64.56 | 54.22 | 16.28
Statistical Analysis 1: Comparison: Group 1; secukinumab 300 mg s.c. injection, week 16; Test type: Superiority; p < 0.0001, Regression, Logistic; Statistical analysis (logistic regression) of PASI75 response by visit in treatment period 1 (non-responder imputation); Odds Ratio, log = 9.49, 95% CI 2-sided [3.73 to 24.16]
Statistical Analysis 2: Comparison: Group 2; secukinumab 150 mg s.c. injection, week 16; Test type: Superiority; p = 0.0001, Regression, Logistic; Statistical analysis (logistic regression) of PASI75 response by visit - in treatment period 1 (non-responder imputation); Odds Ratio (OR) = 6.38, 95% CI 2-sided [2.51 to 16.24]

9. Secondary Outcome: Percentage of Patients Achieving a PASI90 Response in the Subgroup of Subjects Who Have ≥3% Skin Involvement With Psoriasis at Week 16
Description: A 90% reduction in the Psoriasis Area and Severity Index score (PASI 90) is above the current benchmark of primary endpoints for most clinical trials with endpoints of psoriasis.
Time Frame: 16 Weeks
Population: Psoriasis Subset: The psoriasis subset comprises patients having Body Surface Area (BSA) >= 3% at baseline
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 79 | 83 | 43
percentage of participants | 49.37 | 36.14 | 9.3
Statistical Analysis 1: Comparison: Group 1; secukinumab 300 mg s.c. injection, week 16; Test type: Superiority; p < .0001, Regression, Logistic; Statistical analysis (logistic regression) of PASI90 response in treatment period 1 (non-responder imputation); Odds Ratio, log = 9.86, 95% CI 2-sided [3.19 to 30.45]
Statistical Analysis 2: Comparison: Group 2; secukinumab 150 mg s.c. injection, week 16; Test type: Superiority; p = 0.0043, Regression, Logistic; Statistical analysis (logistic regression) of PASI90 response in treatment period 1 (non-responder imputation); Odds Ratio (OR) = 5.21, 95% CI 2-sided [1.68 to 16.21]

10. Secondary Outcome: Percentage of Patients Achieving a PASI100 Response in the Subgroup of Subjects Who Have ≥3% Skin Involvement With Psoriasis at Week 16
Description: A 100% reduction in the Psoriasis Area and Severity Index score (PASI 100) is above the current benchmark of primary endpoints for most clinical trials with endpoints of psoriasis.
  Odds ratio, 95% confidence interval for odds ratio, and p-value are from a logistic regression model with treatment (3 treatment groups), methotrexate usage at baseline (yes, no) and body weight (kg) as explanatory variables.
Time Frame: 16 Weeks
Population: Psoriasis Subset: The psoriasis subset comprises patients having Body Surface Area (BSA) >= 3% at baseline
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 79 | 83 | 43
percentage of participants | 25.32 | 18.07 | 2.33
Statistical Analysis 1: Comparison: Group 1; secukinumab 300 mg s.c. injection, week 16; Test type: Superiority; p = 0.0107, Regression, Logistic; Statistical analysis (logistic regression) of PASI100 response by visit in treatment period 1 (non-responder imputation); Odds Ratio, log = 14.38, 95% CI 2-sided [1.86 to 111.53]
Statistical Analysis 2: Comparison: Group 2; secukinumab 150 mg s.c. injection, week 16; Test type: Superiority; p = 0.0307, Regression, Logistic; Statistical analysis (logistic regression) of PAS100 response by in treatment period 1 (non-responder imputation); Odds Ratio (OR) = 9.82, 95% CI 2-sided [1.24 to 77.90]

11. Secondary Outcome: Change From Baseline to Week 16 in DAS28-CRP
Description: DAS-CRP uses the C-Reactive Protein (CRP) value. Disease Activity Score (DAS28-CRP) values range from 2.0 to 10.0 while higher values mean a higher disease activity. A DAS28-CRP below the value of 2.6 is interpreted as Remission. DAS28-CRP uses 28 different joints for its calculation: proximal interphalangeal joints (10 joints) metacarpophalangeal joints (10) wrists (2) elbows (2) shoulders (2) knees (2) With the above mentioned parameters.
  Least squares mean (LSM), Least squares mean (LSM) treatment difference, 95% confidence interval (CI) for treatment difference, and p-values are from an analysis of covariance (ANCOVA) model with treatment (3 treatment groups), baseline DAS28-CRP score, methotrexate usage at baseline (yes, no), and body weight(kg) as explanatory variables.
Time Frame: baseline, 16 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 103 | 103 | 52
scores on a scale | -1.39 (0.120) | -1.18 (0.125) | -0.35 (0.170)
Statistical Analysis 1: Comparison: Group 1; secukinumab 300mg s.c. injection, 16 weeks; Test type: Superiority; p < .0001, ANCOVA; Statistical analysis (ANCOVA) of change from baseline in DAS28-CRP score in treatment period 1 (LOCF); LS Mean of Treatment Difference = -1.05, 95% CI 2-sided [-1.45 to -0.65]; Standard Error of Treatment Difference 0.203
Statistical Analysis 2: Comparison: Group 2; secukinumab 150 mg s.c. injection; Test type: Superiority; p < .0001, ANCOVA; Statistical analysis (ANCOVA) of change from baseline in DAS28-CRP score in treatment period 1 (LOCF); LS Means of Treatment Difference = -0.83, 95% CI 2-sided [-1.24 to -0.43]; LS Mean of Treatment Difference 0.207

12. Secondary Outcome: Change From Baseline to Week 16 in HAQ-DI
Description: The Health assessment questionnaire disability index (HAQ-DI) is 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0 (no difficulty), to 3 (inability to perform a task in that area). The average score across the functional areas yields an overall HAQ score which ranges from 0 (no disability) to 3 (completely disabled).
Time Frame: 16 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 101 | 101 | 50
scores on a scale | -0.32 [-0.37 to -0.05] | -0.24 [-0.30 to 0.03] | -0.11 [NA to NA] — Placebo not compared to itself. It is below the level of detection
Statistical Analysis 1: Comparison: Group 1; secukinumab 300mg s.c. injection; Test type: Superiority; p = 0.0107, ANCOVA; Statistical analysis (ANCOVA) of change from baseline in HAQ-DI score by in treatment period 1 (LOCF); LS Mean of Treatment Difference = -0.21, 95% CI 2-sided [-0.37 to -0.05]; Standard Error of Treatment Difference 0.081
Statistical Analysis 2: Comparison: Group 2; Test type: Superiority — secukinumab 150 mg s.c. injection; p = 0.1109, ANCOVA; Statistical analysis (ANCOVA) of change from baseline in HAQ-DI score by visit - in treatment period 1 (LOCF); LS Mean Treatment Difference = -0.13, 95% CI 2-sided [-0.30 to 0.03]; Standard Error of Treatment Difference -0.083

13. Other Pre Specified Outcome: Number and Percentage of Patients With ACR20 Response by Visit - in Entire Treatment Period (up to Week 52) (Non-responder Imputation)
Description: Exploratory
  The ACR20 is a composite measure defined as both improvement of 20% in the number of tender and number of swollen joints, and a 20% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [most often Health Assessment Questionnaire (HAQ)], visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP)
Time Frame: up to 52 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Groups:
- Group 2: secukinumab 150 mg s.c. injection (R) Responders
- Group 3: secukinumab 150 mg s.c. injection (NR) Non-responders
- Group 4: Any Secukinumab 150mg
- Group 5: Placebo s.c. injection 300mg
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 103 | 50 | 42 | 103 | 52
percentage of participants
  week 1: number analyzed (Participants) | 18 | 4 | 2 | 6 | 1
  week 1 | 17.48 | 8.00 | 4.76 | 5.83 | 1.92
  week 16: number analyzed (Participants) | 53 | 36 | 2 | 38 | 12
  week 16 | 51.46 | 72.00 | 4.76 | 36.89 | 23.08
  week 52: number analyzed (Participants) | 49 | 34 | 12 | 46 | 22
  week 52 | 47.57 | 68.00 | 28.57 | 44.66 | 42.31

14. Other Pre Specified Outcome: Number and Percentage of Patients With ACR50, ACR70 Response by Visit - in Entire Treatment Period (up to Week 52) (Non-responder Imputation)
Description: Exploratory
Time Frame: up to 52 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 103 | 50 | 42 | 103 | 52
percentage of participants
  ACR50 - week 1: number analyzed (Participants) | 3 | 0 | 1 | 1 | 0
  ACR50 - week 1 | 2.91 |  | 2.38 | .97 |
  ACR70 - week 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  ACR50 - week 16: number analyzed (Participants) | 29 | 23 | 2 | 25 | 3
  ACR50 - week 16 | 28.16 | 46.00 | 4.76 | 24.27 | 5.77
  ACR70 - week 16: number analyzed (Participants) | 18 | 11 | 0 | 11 | 1
  ACR70 - week 16 | 17.48 | 22.00 |  | 10.68 | 1.92
  ACR50 - week 52: number analyzed (Participants) | 33 | 24 | 6 | 30 | 9
  ACR50 - week 52 | 32.04 | 48.00 | 14.29 | 29.13 | 17.31
  ACR70 - week 52: number analyzed (Participants) | 22 | 14 | 2 | 16 | 3
  ACR70 - week 52 | 21.36 | 28.00 | 4.76 | 15.53 | 5.77

15. Other Pre Specified Outcome: Number and Percentage of Patients With Presence of Dactylitis by Visit - in Entire Treatment Period (up to Week 52) (Non-responder Imputation)
Description: Exploratory
Time Frame: up to 52 weeks
Population: Dactylitis Subset
  The Dactylitis Subset comprised patients who had LDI ≥1 at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 103 | 50 | 42 | 103 | 52
percentage of participants
  week 1: number analyzed (Participants) | 44 | 21 | 15 | 42 | 17
  week 1 | 42.72 | 42.00 | 35.71 | 40.78 | 32.69
  week 16: number analyzed (Participants) | 26 | 12 | 11 | 23 | 15
  week 16 | 25.24 | 24.00 | 26.19 | 22.33 | 28.85
  week 52: number analyzed (Participants) | 11 | 3 | 5 | 8 | 5
  week 52 | 10.68 | 6.00 | 11.90 | 7.77 | 9.62

16. Other Pre Specified Outcome: Number and Percentage of Patients With Presence of Enthesitis by Visit - in Entire Treatment Period (up to Week 52) (Non-responder Imputation)
Description: Exploratory
Time Frame: up to 52 weeks
Population: Leeds Enthesitis Index (LEI) Subset:
  The LEI Subset comprised patients who had LEI ≥1 at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 66 | 33 | 27 | 67 | 34
percentage of participants
  week 1: number analyzed (Participants) | 56 | 22 | 24 | 52 | 27
  week 1 | 84.85 | 66.67 | 88.89 | 77.61 | 79.41
  week 16: number analyzed (Participants) | 37 | 8 | 21 | 35 | 28
  week 16 | 56.06 | 24.24 | 77.78 | 52.24 | 82.35
  week 52: number analyzed (Participants) | 35 | 12 | 18 | 36 | 21
  week 52 | 53.03 | 36.36 | 66.67 | 53.73 | 61.76

17. Other Pre Specified Outcome: Number and Percentage of Patients With Minimal Disease Activity Response by Visit in Entire Treatment Period (up to Week 52) (Non-responder Imputation)
Description: Exploratory
Time Frame: up to 52 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 103 | 50 | 42 | 103 | 52
percentage of participants
  week 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  week 1 | 0.97 |  |  |  |
  week 16: number analyzed (Participants) | 24 | 23 | 7 | 30 | 9
  week 16 | 36.36 | 69.70 | 25.93 | 44.78 | 26.47
  week 52: number analyzed (Participants) | 27 | 21 | 6 | 27 | 2
  week 52 | 26.21 | 42.00 | 14.29 | 26.21 | 3.85

18. Other Pre Specified Outcome: Number and Percentage of Patients With PASI75, PASI90 and PASI100 Response by Visit - in Entire Treatment Period (up to Week 52) (Non-responder Imputation)
Description: Exploratory
Time Frame: up to 52 weeks
Population: Psoriasis subset
  The psoriasis subset comprises patients having Body Surface Area (BSA) >= 3% at baseline
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 79 | 40 | 34 | 83 | 43
percentage of participants
  PASI75 - week 1: number analyzed (Participants) | 7 | 3 | 4 | 7 | 2
  PASI75 - week 1 | 8.86 | 7.5 | 11.76 | 8.43 | 4.65
  PASI90 - week 1: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1
  PASI90 - week 1 | 1.27 |  | 2.94 | 1.2 | 1
  PASI100 - week 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  PASI100 - week 1 |  |  |  |  | 2.33
  PASI75 - week 16: number analyzed (Participants) | 51 | 32 | 13 | 45 | 7
  PASI75 - week 16 | 64.56 | 80.00 | 38.24 | 54.22 | 16.28
  PASI90 - week 16: number analyzed (Participants) | 39 | 24 | 6 | 30 | 4
  PASI90 - week 16 | 49.37 | 60.00 | 17.65 | 36.14 | 9.30
  PASI100 - week 16: number analyzed (Participants) | 20 | 15 | 0 | 15 | 1
  PASI100 - week 16 | 25.32 | 37.50 |  | 18.07 | 2.33
  PASI75 - week 52: number analyzed (Participants) | 53 | 31 | 18 | 49 | 23
  PASI75 - week 52 | 67.09 | 77.50 | 52.94 | 59.04 | 53.49
  PASI90- week 52: number analyzed (Participants) | 38 | 27 | 12 | 39 | 19
  PASI90- week 52 | 48.10 | 67.50 | 35.29 | 46.99 | 44.19
  PASI100 - week 52: number analyzed (Participants) | 25 | 22 | 9 | 31 | 14
  PASI100 - week 52 | 31.65 | 55.00 | 26.47 | 37.35 | 32.56

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from first dose of study treatment until end of study treatment up to maximum duration of 52 weeks plus 12 weeks follow up
Description: An AE is any untoward sign or symptom that occurs in >=5% of participants during study treatment.
  AEs were counted based on the last actual dose received prior to onset of the AE. The secukinumab 300mg group included patients who received secukinumab 300mg for the entire study and those who switched to secukinumab 300mg in Treatment Period 2
Groups:
- Secukinumab 300mg: Secukinumab 300mg
- Secukinumab 150mg: Secukinumab 150mg
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/191 | 0/103 | 1/52
Serious Adverse Events (participants affected / at risk) | 15/191 | 4/103 | 3/52
Other Adverse Events (participants affected / at risk) | 66/191 | 35/103 | 12/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300mg (N=191) | Secukinumab 150mg (N=103) | Placebo (N=52)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Bursitis infective (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Intestinal sepsis (Infections and infestations) | 1 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pubic pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral cyst (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0
Device loosening (Product Issues) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300mg (N=191) | Secukinumab 150mg (N=103) | Placebo (N=52)
Diarrhoea (Gastrointestinal disorders) | 11 | 7 | 2
Bronchitis (Infections and infestations) | 10 | 1 | 1
Nasopharyngitis (Infections and infestations) | 6 | 6 | 1
Sinusitis (Infections and infestations) | 8 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 26 | 6 | 1
Urinary tract infection (Infections and infestations) | 10 | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 8 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 5 | 3
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 3 | 6 | 0
Hypertension (Vascular disorders) | 8 | 6 | 0

LIMITATIONS AND CAVEATS:
Period 2 (week 16 up to 52 weeks) contained only exploratory outcomes. AEs are presented cumulitively

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-12-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT02798211/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT02798211/SAP_001.pdf